CLINICAL TRIAL: NCT00005410
Title: Epidemiology of Coronary Heart Disease in Blacks
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4328; R03HL047208 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease; Myocardial Infarction
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Myocardial Infarction

SUMMARY:
To conduct an analysis of the epidemiology of coronary heart disease (CHD) in Blacks using data collected from the 'Survival and Ventricular Enlargement (SAVE) Following Myocardial Infarction' study.

DETAILED DESCRIPTION:
BACKGROUND:

Ample data now exist to dispel the prevailing clinical impression that coronary heart disease (CHD) occurs infrequently in United States Blacks. It is well known that CHD is the leading cause of death among United States Blacks. Among patients with acute myocardial infarction who often present with typical ischemic chest pain, it has been shown that Blacks present more often without chest pain when compared to whites and Hispanics. In addition, more than 25 percent of the myocardial infarction patients have unrecognized infarctions. Morbidity and mortality associated with angina pectoris, cardiovascular disease, and myocardial infarction occurs in United States Blacks at rates which are at least comparable to their white counterparts. Yet, there are limited epidemiological studies designed to identify the determinants of CHD in the Black population.

The patients were originally screened to participate in a multicenter clinical trial on 'Survival and Ventricular Enlargement (SAVE) Following Myocardial Infarction.' Only 28 patients out of 599 screened subjects were eligible for the SAVE study. The baseline data obtained from the 599 screened subjects comprised the database.

DESIGN NARRATIVE:

Data analysis was performed to: determine the prevalence of coronary heart disease in Blacks presenting with chest pain; identify the correlates of CHD in Blacks; determine the sensitivity and specificity of a Rose questionnaire angina in Blacks; determine the association between the Rose questionnaire angina and CHD manifestations in Blacks, and identify predictive and causal models of CHD.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-06; Study Completion 1993-05 (Actual)

REFERENCES:
- [Background] Peniston RL, Adams-Campbell L, Fletcher JW, Williams EC, Murigande C, Mensah E, Crittenden MD, Diggs JA. Coronary arteriographic findings in black patients and risk markers for coronary artery disease. Am Heart J. 1994 Mar;127(3):552-9. doi: 10.1016/0002-8703(94)90662-9. PMID 8122601
- [Background] Adams-Campbell LL, Peniston RL, Kim KS, Mensah E. Body mass index and coronary artery disease in African-Americans. Obes Res. 1995 May;3(3):215-9. doi: 10.1002/j.1550-8528.1995.tb00141.x. PMID 7627769